CLINICAL TRIAL: NCT04701086
Title: A 3-month, Prospective, Multicentre, Investigator-masked, Parallel-group, Active-controlled, Randomised, Non-inferiority Study to Compare the Efficacy & Tolerability of CATIONORM PRO® & VISMED® in Patients With Mod-to-severe Dry Eye Disease
Brief Title: 3 Month Study of Cationorm Pro Versus Vismed in Adults With Dry Eye Disease Related to Keratitis or Keratoconjunctivitis
Acronym: PROSIKA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Santen SAS (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RE-010-2020-SA
Record Dates: First submitted 2021-01-05; First posted 2021-01-08 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Dry Eye Syndromes
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Intervention Model Description: PROSPECTIVE, MULTICENTRE, INVESTIGATOR-MASKED, PARALLEL-GROUP, ACTIVE-CONTROLLED, RANDOMISED, NON-INFERIORITY STUDY
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Investigator Masked, unmasked Pharmacist
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cationorm Pro (Experimental): Cationorm Pro is an ophthalmic sterile unpreserved eye drops emulsion (N=40) Posology: One Drop in each eye 4 times daily for 84 days
  Interventions: Device: Cationorm Pro
- Vismed (Active Comparator): HA 0.18% hyaluronic solution (N40) Posology: One Drop in each eye 4 times daily for 84 days
  Interventions: Device: Vismed

INTERVENTIONS:
Device: Cationorm Pro — Eye Drops
  Other Names: Ocutears Pro+
  Arms: Cationorm Pro
Device: Vismed — Eye Drops
  Arms: Vismed

SUMMARY:
This study is a prospective, multicentre, parallel-group, active-controlled, non-inferiority study conducted in adult patients with moderate-to-severe dry eye disease (DED) related to keratitis or keratoconjunctivitis. This study is to be conducted in France, Poland and Spain.

The patients will be randomised to receive Cationorm Pro® or the reference treatment, VISMED® (ratio 1:1) in an investigator-masked fashion

DETAILED DESCRIPTION:
Primary:

• To compare the ocular efficacy of Cationorm Pro® with that of VISMED® in patients with moderate to severe DED related to keratitis or keratoconjunctivitis after a 4-week treatment period (Day 28).

Secondary:

To compare the ocular efficacy of Cationorm Pro® with that of VISMED® in patients with moderate to severe DED related to keratitis or keratoconjunctivitis over a 12-week treatment period To evaluate the ocular tolerability and safety of Cationorm Pro® versus VISMED® in patients with moderate to severe DED related to keratitis or keratoconjunctivitis throughout the duration of treatment

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patient aged 18 years or above.
2. Patient using artificial tears for at least 3 months prior to the Screening visit.
3. Patient experiencing at least 2 symptoms of ocular discomfort rated ≥23 mm on the 0 to 100 mm visual analogue scale (VAS) (among itching, eye dryness, sticky feeling, photophobia, pain, burning or stinging, sandy feeling or grittiness, or foreign body sensation) at Screening and Baseline visits.
4. OSS score (sum of nasal and temporal interpalpebral conjunctival and corneal vital staining) ≥4 and ≤9 on a modified Oxford scale at Screening and Baseline visits in at least one eye.
5. TBUT of ≤10 seconds at Screening and Baseline visits and/or Schirmer's tear test of ≥3 and ≤9 mm/5 min at Screening visit in the same eye that fulfil inclusion criteria #4.
6. The patient has signed and dated a written informed consent form prior to the initiation of any study procedures.

   -

Exclusion Criteria:

the study: Ocular

1. CFS score ≥4 on a modified Oxford scale
2. Ocular hypertension or glaucoma requiring IOP-lowering medication(s)
3. History of ocular trauma, infection or ocular inflammatory condition within the last 3 months before the screening visit.
4. Severe blepharitis and/or severe meibomian gland disease
5. Filamentary keratitis
6. Any ocular surface anomaly not related to DED
7. Active ocular infection or history of ocular allergy or ocular herpes
8. Patient with only one sighted eye or with a best corrected distance visual acuity ≤1/10
9. Use of any topical ocular treatment other than study device during the study (all non-study topical ocular treatment(s) must be stopped at the screening visit)
10. Onset of lid hygiene (whatever the method) less than 2 months before the Screening visit
11. Use of topical corticosteroids one month before the Screening Visit
12. Use of isotretinoin, ciclosporin, tacrolimus, sirolimus, pimecrolimus or ocular cauterisation procedures 2 months before the screening visit and throughout the study
13. Use of VISMED® within 6 weeks prior to the screening visit
14. Refractive surgery (e.g. LASIK, LASEK, PRK) within 6 months and/or any other ocular laser/surgery within 3 months prior to the screening visit and during the study
15. Insertion of temporary punctal plug(s) within 2 months prior to the Screening visit or permanent occlusion of lacrimal puncta on one or both sides
16. Known hypersensitivity to any of the components of the study device or investigational products Non-ocular
17. History of severe systemic allergy
18. Systemic disease not stabilised within 1 month prior to the screening visit (e.g. diabetes with glycaemia out of range, thyroid dysfunction) or judged by the investigator to be incompatible with the conduct of the study procedures or the interpretation of the study results
19. Any change of systemic concomitant medication within the month before the screening visit or planned change during the study period, except paracetamol
20. Pregnancy or lactation at the screening and/or Baseline visit.
21. Women of childbearing potential not using a medically acceptable, highly effective method of birth control (such as hormonal implants, injectable or oral contraceptives together with condoms, some intrauterine devices, sexual abstinence or vasectomised partner) from the Baseline visit throughout the conduct of the study treatment periods and up to 2 weeks after the study end. Post-menopausal women (two years without menstruation) do not need to use any method of birth control.
22. Participation in a clinical trial with an investigational substance within the past 30 days prior to Baseline visit.
23. Participation in another clinical study at the same time as the present study. -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2021-09-30 (Actual); Primary Completion 2025-04-28 (Actual); Study Completion 2025-04-28 (Actual)

PRIMARY OUTCOMES:
Change of ocular surface staining (OSS) score between baseline and Day 28. | Between Baseline and day 28
  The primary endpoint of the study is the difference between patients treated with Cationorm Pro® and patients treated with VISMED® in the change of ocular surface staining (OSS) score between baseline and D28.
  An OSS higher than 0 is considered to be abnormal and may be a sign of KCS. But scores of 1 or 2 can also represent a late staining artifact if interpretation of the fluorescein corneal staining pattern is delayed beyond 8 minutes. Because this could lead to a high level of misclassification, an abnormal OSS is defined as being a score of 3 or above.

SECONDARY OUTCOMES:
Change of ocular surface staining (OSS) score between baseline and Day 84 | between baseline and Day 14 and between baseline and Day 84
  The difference between patients treated with Cationorm Pro® and patients treated with VISMED® in change of OSS score between baseline and Day 84.
  An OSS higher than 0 is considered to be abnormal and may be a sign of KCS. But scores of 1 or 2 can also represent a late staining artifact if interpretation of the fluorescein corneal staining pattern is delayed beyond 8 minutes. Because this could lead to a high level of misclassification, an abnormal OSS is defined as being a score of 3 or above.
The change of ocular stainings (corneal fluorescein staining (CFS) and conjunctival staining) between baseline and Day 28 and between baseline and Day 84 | between baseline and Day 28 and between baseline and Day 84
  The difference between patients treated with Cationorm Pro® and patients treated with VISMED® in change of ocular stainings (corneal fluorescein staining (CFS) and conjunctival staining)
  Staining using fluorescein will be graded using the modified Oxford scale (7-point ordinal scale, score 0, 0.5, and 1 to 5 per area [cornea + nasal and temporal conjunctiva]) for cornea and conjunctiva separately, On this modified scale, the score 0 corresponds to no staining dots and the score 0.5 corresponds to one staining dot per area. A CFS grade of 0 represents complete corneal clearing.
The change of ocular discomfort symptoms on Visual Analogue Scale | between baseline and Day 28 and between baseline and Day 84
  The difference between patients treated with Cationorm Pro® and patients treated with VISMED® in the change of ocular discomfort symptoms according to the Visual Analogue Scale (VAS)
  Patient experiencing at least 2 symptoms of ocular discomfort rated ≥23 mm on the 0 to 100 mm visual analogue scale (VAS) (among itching, eye dryness, sticky feeling, photophobia, pain, burning or stinging, sandy feeling or grittiness, or foreign body sensation) at Screening and Baseline visits.
The change tear breakup time (TBUT) | between baseline and Day 28 and between baseline and Day 84
  The difference between patients treated with Cationorm Pro® and patients treated with VISMED® in the change of tear breakup time (TBUT)
  Generally, >10 seconds is thought to be normal,(10, 11, 12) 5 to 10 seconds, marginal, and < 5 seconds is considered low. A short tear break-up time is a sign of a poor tear film and the longer it takes the more stable the tear film.
The change in Schirmer's tear test | between baseline and Day 28 and between baseline and Day 84
  The difference between patients treated with Cationorm Pro® and patients treated with VISMED® in the change of Schirmer's tear test
  Healthy eyes are considered to leave each strip of paper containing more than 10 millimeters of moisture. Less than 10 millimeters of moisture indicates probable dry eye syndrome
The secondary endpoints are the difference between patients treated with Cationorm Pro® and patients treated with VISMED® in the change of overall efficacy evaluation of the investigator | after 12 weeks of treatment (84 days)
  The study investigator at each centre will conduct an overall assessment of the effect of the study device on improvement in the patients DED using the following rating scale:
  0 = Unsatisfactory
  1. = Not very satisfactory
  2. = Satisfactory
  3. = Very satisfactory
The difference between patients treated with Cationorm Pro® and patients treated with VISMED® in the change of subjective assessments evaluation by the patient. | between baseline and Day 84
  The patient will rate his global evaluation of efficacy using the same rating scale as the Investigator.
  A subjective assessment is completed of the effect of the study device on improvement in their DED using the following rating scale:
  0 = Unsatisfactory
  1. = Not very satisfactory
  2. = Satisfactory
  3. = Very satisfactory

CONTACTS AND LOCATIONS:
Locations (8):
- CHRU Bretonneau, Tours, France
- Poland (3):
  - Gabinet Okulistyczny, Bielsko-Biala
  - 5th MILITARY CLINICAL HOSPITAL IN KRAKOW, Krakow
  - Szpital SW. Rozy, Krakow
- Spain (4):
  - Centro de Oftalmologia Barraquer, Barcelona
  - Hospital Clinic of Barcelona, Barcelona
  - Hospital Unniversitario Donostia, Donostia / San Sebastian
  - El Instituto Ofalmológico Quirónsalud Zaragoza, Zaragoza

IPD SHARING:
Plan to Share IPD: No